CLINICAL TRIAL: NCT07293780
Title: The Effect of Transcranial Magnetic Stimulation Applied to the Primary Motor Cortex and Anterior Cingulate Cortex on Refractory Neuropathic Pain in Spinal Cord Injury
Brief Title: Effect of TMS on Neuropathic Pain for Patients With Sci
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-102
Record Dates: First submitted 2025-11-13; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active rTMS primer motor cortex (Active Comparator)
  Interventions: Device: active TMS
- rTMS anterior cingulate gyrus (Experimental)
  Interventions: Device: active TMS
- sham rTMS primer motor cortex (Sham Comparator)
  Interventions: Device: sham TMS

INTERVENTIONS:
Device: active TMS — Patients in the active or sham primary motor cortex rTMS group will receive active or sham rTMS at 5 Hz targeting the M1 area of the lower extremity motor area under medical supervision for a total of 10 sessions over 2 weeks. Patients in the active anterior cingulate cortex rTMS group will also receive active 5 Hz rTMS targeting the anterior cingulate cortex for a total of 10 sessions over 2 weeks under medical supervision.
  Arms: active rTMS primer motor cortex; rTMS anterior cingulate gyrus
Device: sham TMS — Patients in the active or sham primary motor cortex rTMS group will receive active or sham rTMS at 5 Hz targeting the M1 area of the lower extremity motor area under medical supervision for a total of 10 sessions over 2 weeks. Patients in the active anterior cingulate cortex rTMS group will also receive active 5 Hz rTMS targeting the anterior cingulate cortex for a total of 10 sessions over 2 weeks under medical supervision.
  Arms: sham rTMS primer motor cortex

SUMMARY:
The aim of this study is to evaluate the efficacy of rTMS targeting the anterior cingulate cortex, another stimulation site that may be effective in the treatment of neuropathic pain, and to compare it with motor cortex stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients for whom at least 12 months have passed since the date of the event
2. Patients who meet the International Pain Working Group's criteria for central neuropathic pain below the level of the lesion and who have had pain for at least 6 months
3. Patients aged 18-65
4. Pain not attributable to other causes such as rheumatological diseases or diabetes
5. Patients with VAS > 4 despite maximum dose of pharmacological agents (anticonvulsants, antidepressants, narcotics), exercise and physical therapy agents, taking into account renal function tests and other comorbidities

Exclusion Criteria:

1. History of epilepsy
2. Metallic implant in the scalp
3. Cochlear implant
4. Spinal cord stimulator
5. Pacemaker
6. Presence of psychiatric illness
7. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | first day of treatment, at the end of treatment (at 2nd week), 4 week after end of treatment, 12 week after end of treatment
  The assessment of pain using a 10 cm visual analogue scale (VAS), separately for daytime and night-time. The assessment will be conducted on a scale of "0 = no pain" to "10 = the most severe pain imaginable".

SECONDARY OUTCOMES:
neuropathic pain scale | first day of treatment, at the end of treatment (at 2nd week), 4 week after end of treatment, 12 week after end of treatment
Beck Depression Scale | first day of treatment, at the end of treatment (at 2nd week), 4 week after end of treatment, 12 week after end of treatment
5-point Likert scale | first day of treatment, at the end of treatment (at 2nd week), 4 week after end of treatment, 12 week after end of treatment
  It is a 5-point Likert scale to be used for assessing patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Etlik City Hospital, Ankara, Yenimahalle
  - Gaziler Physical Therapy and Rehabilitation Training and Research Hospital, Ankara, Çankaya